CLINICAL TRIAL: NCT00654940
Title: Methodology Study To Assess The Ability Of A Randomized, Double-Blind, Placebo-Controlled, Two Period Crossover Study To Detect The Effect Of Pregabalin In Post-Traumatic Neuropathic Pain Patients
Brief Title: A Study To Assess The Ability Of A Crossover Study Design To Detect The Efficacy Of Pregabalin In Post-Traumatic Neuropathic Pain Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: A0081187
Record Dates: First submitted 2008-04-03; First posted 2008-04-09 (Estimated); Results first posted 2010-02-24 (Estimated); Last update posted 2021-02-09 (Actual); Status verified 2010-02

CONDITIONS: Nerve Pain
MeSH Terms: conditions — Neuralgia | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator)
  Interventions: Drug: Pregabalin (Lyrica)
- B (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pregabalin (Lyrica) — Oral, 75mg or 150mg capsules, BID
  Arms: A
Drug: Placebo — Oral, matched capsules, BID
  Arms: B

SUMMARY:
The purpose of this study is to assess whether a cross-over type study design in post-traumatic neuropathic patients can be used to assess the activity of potential analgesic agents

DETAILED DESCRIPTION:
Methodology study to evaluate a cross-over study design in post-traumatic neuropathic pain patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients require a diagnosis of post-traumatic peripheral neuropathic pain (NeP), including post-surgical NeP and NeP due to peripheral nerve injury, which has lasted at least 3 months following the traumatic event.
* Patients during the screening week must have completed ≥ 4 daily pain scores and have an average daily pain score ≥ 4.
* Female patients of childbearing potential must have a negative urine pregnancy test at Screening and be practicing an acceptable form of contraception.

Exclusion Criteria:

* Patients with neuropathic pain (NeP) that is not due to trauma; e.g. patients with trigeminal neuralgia, central pain, complex region pain syndrome type I, phantom limb pain, radiculopathy, painful diabetic neuropathy or post-herpetic neuralgia or patients with any other co-existing pain which cannot be differentiate from NeP of peripheral origin.
* Patients who have previously failed to respond to pregabalin at a total daily dose of equal to or greater than 300 mg or are intolerant to those doses.
* Patients who have previously failed to respond to gabapentin at a total daily dose of equal to or greater than 1800 mg.
* Patients with any type or history of malignancy, except either where there has been no ongoing treatment for at least 6 months or all basal cell carcinomas; all patients with a history of brain or spinal tumors will be excluded.
* Patients who currently have ongoing litigation related to any injury affecting their pain symptomatology.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2008-05; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (5):
- Canada (3):
  - Pfizer Investigational Site, Calgary, Alberta
  - Pfizer Investigational Site, Hamilton, Ontario
  - Pfizer Investigational Site, Sarnia, Ontario
- Sweden (2):
  - Pfizer Investigational Site, Jönköping
  - Pfizer Investigational Site, Linköping

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081187&StudyName=A%20Study%20To%20Assess%20The%20Ability%20Of%20A%20Crossover%20Study%20Design%20To%20Measure%20The%20Activity%20Of%20Pregabalin%20In%20Post-Traumatic%20Neuropathic%20Pain%20P

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects participated in the study between 05 May 2008 and 10 February 2009.
Pre-assignment Details: Subjects meeting entry criteria entered into a 1-week screening period to monitor daily pain scores and activity levels. If pain severity met inclusion criteria subjects could enter the double-blind part of the study and were randomized to 1 of 2 treatment sequence crossovers (pregabalin/placebo or placebo/pregabalin).
Groups:
- Pregabalin First Then Placebo: Pregabalin: Day 1: 75 mg in the evening, Days 2 & 3: 150 mg/day, Day 4: 225 mg/day, Days 5 to 14: 300 mg/day, Day 15: 150 mg in the morning. Twice daily (BID) dosing on Days 2-14. Placebo: Day 1 in the evening, Days 2-14 BID, Day 15 in the morning.
- Placebo First Then Pregabalin: Placebo: Day 1 in the evening, Days 2-14 BID, Day 15 in the morning. Pregabalin: Day 1: 75 mg in the evening, Days 2 & 3: 150 mg/day, Day 4: 225 mg/day, Days 5 to 14: 300 mg/day, Day 15: 150 mg in the morning. Twice daily (BID) dosing on Days 2-14.
Period: Period 1
Arm/Group | Pregabalin First Then Placebo | Placebo First Then Pregabalin
Started | 13 (Assigned to study treatment.) | 12 (Assigned to study treatment.)
Received Study Treatment | 12 | 12
Completed | 12 | 11
Not Completed | 1 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Intolerable Pain Level | 1 | 0
Period: Washout Period of 2 Weeks
Arm/Group | Pregabalin First Then Placebo | Placebo First Then Pregabalin
Started | 12 | 11
Completed | 12 | 11
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Pregabalin First Then Placebo | Placebo First Then Pregabalin
Started | 12 | 11
Completed | 12 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Pregabalin Then Placebo: Pregabalin: Day 1: 75 mg in the evening, Days 2 & 3: 150 mg/day, Day 4: 225 mg/day, Days 5 to 14: 300 mg/day, Day 15: 150 mg in the morning. BID dosing Days 2-14. Placebo: Day 1 in the evening, Days 2 to 14 BID, Day 15 in the morning.
- Placebo Then Pregabalin: Placebo: Day 1 in the evening, Days 2 to 14 BID, Day 15 in the morning. Pregabalin: Day 1: 75 mg in the evening, Days 2 & 3: 150 mg/day, Day 4: 225 mg/day, Days 5 to 14: 300 mg/day, Day 15: 150 mg in the morning. BID dosing Days 2-14.
- Total: Total of all reporting groups
Arm/Group | Pregabalin Then Placebo | Placebo Then Pregabalin | Total
Number analyzed (Participants) | 13 | 12 | 25
Age, Customized [Number; unit: years]
  18 - 44 years | 4 (0) | 3 (0) | 7 (0)
  45 - 64 years | 5 (16.7) | 8 (11.8) | 13
  >=65 years | 4 (0) | 1 (0) | 5 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Treatment Week 2 in Daily Pain Rating Scale
Description: Daily Pain Rating Scale by treatment and sequence using an 11-point Likert scale: range 0 (no pain) to 10 (worst possible pain) over the past 24 hours. Self-assessment was performed daily on rising from bed (for the final time in the case of interrupted sleep). Average daily pain score: mean of the previous 7 days daily pain scores. Baseline was defined as the mean of the last 7 pre-treatment pain scores for each period. End of treatment was defined as the mean of the last 7 on treatment pain scores for each period.
Time Frame: Week 0 to Week 2, Week 4 to Week 6 (Baseline to Week 2 [End of Treatment] for each treatment period)
Population: Full Analysis Set: (FAS): all subjects randomized who received at least one dose of study drug, regardless of whether they had efficacy data. Baseline is Week 0 and Week 4 for Periods 1 and 2, respectively. Treatment Week 2 is End of Treatment (Week 2 and Week 6) for Periods 1 and 2, respectively.
Measure: Mean (Standard Deviation); unit: scores on scale
Groups:
- Period 1: Pregabalin; Period 2: Pregabalin: Day 1: 75 mg in the evening, Days 2 & 3: 150 mg/day, Day 4: 225 mg/day, Days 5 to 14: 300 mg/day, Day 15: 150 mg in the morning. BID dosing on Days 2-14.
- Period 1: Placebo; Period 2: Placebo: Day 1 in the evening, Days 2-14 BID, Day 15 in the morning.
Arm/Group | Period 1: Pregabalin | Period 1: Placebo | Period 2: Placebo | Period 2: Pregabalin
Number analyzed (Participants) | 13 | 12 | 12 | 11
scores on scale
  Baseline | 6.03 (1.29) | 5.24 (2.03) | 5.96 (0.88) | 5.31 (1.82)
  Treatment Week 2 | 5.40 (1.34) | 5.08 (2.05) | 6.11 (1.20) | 4.38 (2.02)
  Change from Baseline | -0.63 (1.01) | -0.16 (0.97) | 0.16 (1.07) | -0.93 (1.24)
Statistical Analysis 1: Comparison: Period 1: Pregabalin vs Period 1: Placebo vs Period 2: Placebo vs Period 2: Pregabalin; Treatment comparison of pregabalin - placebo: mixed effects analysis of covariance model fitted on the full analysis set population, accounting for period and treatment effects. Subject was fitted as a random effect, and baseline was fitted as two covariates; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.81, 80% CI [-1.21 to -0.41], Standard Error of Mean 0.305

2. Secondary Outcome: Neuropathic Pain Symptom Inventory (NPSI)
Description: NPSI at end of treatment: 10-item self-administered questionnaire assessing 5 dimensions of pain (burning superficial spontaneous pain, pressing deep spontaneous pain, paroxysmal pain, evoked pain, and paresthesia/dysesthesia). Each item consists of a question about the specific qualities of pain and an 11-point numerical scale range: 0 (absence of pain) to 10 (maximum intensity imaginable), and 2 temporal items related to spontaneous and paroxysmal pain. Maximum total score possible = 100.
Time Frame: Week 0 to Week 2, Week 4 to Week 6 (Baseline to End of Treatment in Treatment Periods 1 and 2)
Population: FAS. Weeks 0 and 4 are baseline for Periods 1 and 2, respectively. Weeks 2 and 6 are End of Treatment for Periods 1 and 2, respectively.
Measure: Mean (Standard Deviation); unit: scores on scale
Groups:
- Pregabalin/Placebo: Pregabalin Day 1: 75 mg in the evening, Days 2 & 3: 150 mg/day, Day 4: 225 mg/day, Days 5 to 14: 300 mg/day, Day 15: 150 mg in the morning. BID dosing on Days 2-14. Placebo: Day 1 in the evening, Days 2-14 BID, Day 15 in the morning.
- Placebo/Pregabalin: Placebo: Day 1 in the evening, Days 2-14 BID, Day 15 in the morning. Pregabalin Day 1: 75 mg in the evening, Days 2 & 3: 150 mg/day, Day 4: 225 mg/day, Days 5 to 14: 300 mg/day, Day 15: 150 mg in the morning. BID dosing on Days 2-14.
Arm/Group | Pregabalin/Placebo | Placebo/Pregabalin
Number analyzed (Participants) | 13 | 12
scores on scale
  Week 0 (Baseline: Treatment Period 1) | 5.31 (3.50) | 5.25 (2.38)
  Week 2 (End of Treatment: Treatment Period 1) | 5.31 (3.30) | 4.91 (2.30)
  Week 4 (Baseline: Treatment Period 2) | 4.33 (3.14) | 5.27 (2.45)
  Week 6 (End of Treatment: Treatment Period 2) | 4.75 (3.39) | 3.00 (2.24)
Statistical Analysis 1: Comparison: Pregabalin/Placebo vs Placebo/Pregabalin; Neuropathic Pain Symptom Inventory treatment comparison: Pregabalin - Placebo. Total score was analyzed using a mixed effect analysis of covariance model based on the full analysis set (FAS), accounting for period and treatment effects. Subject was fitted as a random effect and baseline was fitted as two covariates; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.52, 80% CI [-3.82 to 2.78], Standard Error of Mean 2.493

3. Secondary Outcome: Subject Activity as Captured by the Actiwatch Score Device: Total Activity Score at End of Treatment
Description: Total activity score: Day (8 am to 8 pm) at end of treatment. Accelerometer measured physical activity by monitoring degree and intensity of body motion. Data is reported as activity counts. Subject activity was collected hourly for the variables: peak, average, and total activity. Higher score indicates greater activity (no activity = 0; total possible score was not defined).
Time Frame: Week 0 to Week 2, Week 4 to Week 6 (Baseline to End of Treatment in Treatment Periods 1 and 2)
Population: FAS; End of Treatment is treatment week 2 (Week 2 and Week 6) for Periods 1 and 2.
Measure: Least Squares Mean (Standard Error); unit: scores on scale
Groups:
- Pregabalin: Day 1: 75 mg in the evening, Days 2 & 3: 150 mg/day, Day 4: 225 mg/day, Days 5 to 14: 300 mg/day, Day 15: 150 mg in the morning. BID dosing on Days 2-14.
- Placebo: Day 1 in the evening, Days 2-14 BID, Day 15 in the morning.
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 24 | 24
scores on scale | 300000 (12000) | 270000 (12000)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Difference in least squares means Pregabalin-Placebo. Model of day (8 am to 8 pm) total activity score at end of treatment. Mixed effects analysis of covariance model was fitted on the full analysis set population, accounting for period and treatment effects. Subject was fitted as a random effect and baseline was fitted as two covariates; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 29000, 80% CI [6100 to 51000], Standard Error of Mean 17000

ADVERSE EVENTS:
Description: Safety analysis set: all randomized subjects who received study medication. Twenty-four (24) subjects received both pregabalin and placebo and were evaluated for adverse events; this includes 12 subjects who started on pregabalin and crossed over to placebo, and 12 subjects who started on placebo and crossed over to pregabalin.
Groups:
- Pregabalin: Day 1: 75 mg in the evening, Days 2 & 3: 150 mg/day, Day 4: 225 mg/day, Days 5 to 14: 300 mg/day, Day 15: 150 mg in the morning. BID dosing Days 2-14.
- Placebo: Day 1 in the evening, Days 2 to 14 BID, Day 15 in the morning.
Arm/Group | Pregabalin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 11/24 | 10/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin (N=24) | Placebo (N=24)
Vertigo (Ear and labyrinth disorders) | 0 | 1
Eye disorder (Eye disorders) | 1 | 0
Vision blurred (Eye disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Dry mouth (Gastrointestinal disorders) | 2 | 1
Hypoaesthesia oral (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 4 | 3
Fatigue (General disorders) | 2 | 1
Influenza like illness (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 1
Therapeutic response unexpected (General disorders) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 1
Increased appetite (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Disturbance in attention (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 6 | 1
Dysgeusia (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 3 | 0
Somnolence (Nervous system disorders) | 3 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Thinking abnormal (Psychiatric disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Diaphragmalgia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1
Hot flush (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.